CLINICAL TRIAL: NCT07229261
Title: MitoQ (Mitoquinol Mesylate) to Ameliorate Vascular Function in Preeclampsia: a Novel Approach
Brief Title: MitoQ to Improve Vascular Funciton in Preeclampsia
Acronym: MAVEN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Jennifer McIntosh, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO00056100
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-07

CONDITIONS: Preeclampsia; Pregnancy
Keywords: pregnancy; preeclampsia; MitoQ; Mitoquinone; Endothelial Function
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Preeclampsia with Severe Features taking Mitoquinol Mesylate (Experimental): Patients allocated to this arm will be inpatients who have preeclampsia with severe features. They will receive 10mg of Mitoquinol Mesylate daily from enrollment until delivery.
  Interventions: Dietary Supplement: Mitoquinol Mesylate
- Preeclampsia with Severe Features taking placebo (Placebo Comparator): Patients allocated to this arm will be inpatients who have preeclampsia with severe features. They will receive Placebo daily from enrollment until delivery.
  Interventions: Other: Placebo
- Preeclampsia without Severe Features taking MitoQ (Experimental): Patients allocated to this arm will be out-patients who have preeclampsia without severe features. They will receive 10mg of Mitoquinol Mesylate daily from enrollment until delivery.
  Interventions: Dietary Supplement: Mitoquinol Mesylate
- Preeclampsia without Severe Features taking placebo (Placebo Comparator): Patients allocated to this arm will be out-patients who have preeclampsia without severe features. They will receive placebo daily from enrollment until delivery.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Mitoquinol Mesylate — Patients randomized to the intervention will receive 10mg of Mitoquinol Mesylate daily from enrollment until delivery.
  Arms: Preeclampsia with Severe Features taking Mitoquinol Mesylate; Preeclampsia without Severe Features taking MitoQ
Other: Placebo — Patients randomized to the placebo groups will take 1 placebo capsule daily until delivery.
  Arms: Preeclampsia with Severe Features taking placebo; Preeclampsia without Severe Features taking placebo

SUMMARY:
Preeclampsia is a leading cause of maternal and neonatal morbidity and mortality. There is a lack of effective therapeutics for prevention or treatment. Our previous ex vivo work demonstrated that mitochondrial-antioxidants can reverse placental microvascular damage. Therefore, this study will evaluate whether MitoQ (Mitoquinol Mesylate, a mitochondrial-antioxidant) has the potential to restore vasodilation, improve placental function, and therefore promote pregnancy prolongation in patients with preeclampsia. This evaluation of clinical data, patient samples, and vascular function studies in patients with preeclampsia could translate into a viable therapeutic option.

DETAILED DESCRIPTION:
Preeclampsia (PreE) impacts ~10% of pregnancies and has severe outcomes both during and after pregnancy. It is a leading cause of pregnancy-related deaths, and has long term cardiovascular consequences for maternal and child health. Despite advances in our understanding of preeclampsia over the past 50 years, the underlying unifying mechanism causing preeclampsia remains elusive. This critical gap not only encompasses lack of understanding of the pathophysiology, but it also includes a lack of therapeutics for prevention or treatment. Success in this study could translate into a clinical trial that could finally offer a treatment for PreE.

We have recently demonstrated that endothelial function in the human placental microcirculation is impacted by excess reactive oxygen and nitrogen species (ROS, RNS) from the mitochondria (MT), which in preeclampsia, impairs vasodilation. Excess ROS causes decreased nitric oxide (NO) bioavailability, increased lipid peroxidation, uncoupled eNOS, peroxynitrite, and exacerbates MT dysfunction and MT DNA damage via alterations in NO. Microvascular function can be improved by mechanisms that rebalance the oxidative stress response. We have shown that MitoTempol, a MT antioxidant, improves vasodilation. Moreover, we have shown that a major part of the cycle of excessive oxidative stress is caused by MT DNA damage and subsequent activation of toll like receptor 9 (TLR9), and that inhibiting TLR9 prevents this dysfunction. The finding that MT antioxidants given ex-vivo can reverse placental vascular damage after delivery gives promise that treatment of patients during pregnancy could restore vasodilation and allow for safer prolongation of pregnancy.

MitoQ (Mitoquinol Mesylate) is a nutritional supplement, and mitochondrial antioxidant. MitoQ has been extensively studied pre- clinically in cell-culture, and pregnant mouse, rat, and sheep models of PreE or oxidative stress and demonstrated beneficial fetal results. It has been used in clinical trials for heart failure, hepatitis C, Parkinson's, and multiple sclerosis with doses from 10mg to 80mg per day.

Overall Hypothesis: We hypothesize that MitoQ (Mitoquinol Mesylate)-treated preeclampsia patients will have improved brachial artery flow-mediated dilation (FMD) and laser Doppler flowmetry assessments of the cutaneous microvasculature, and that placental endothelial function in micro-vessels and placental pathology will be improved in treated patients. To demonstrate this, we will enroll two pilot human cohorts- one of admitted patients with preeclampsia with severe features who will either continue standard in-patient clinical care or be supplemented daily with MitoQ (Mitoquinol Mesylate) and a second outpatient cohort of patients with preeclampsia without severe features who will received standard outpatient care or be supplemented daily with MitoQ

Aim: Test whether with MitoQ (Mitoquinol Mesylate) treatment in preeclamptic patients improves endothelial function Hypothesis: MitoQ (Mitoquinol Mesylate)-treated patients will have improved brachial artery FMD and laser Doppler flowmetry assessments of the cutaneous microvasculature and placental endothelial function in micro-vessels and placental pathology will be improved in treated patients.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient Cohort

  * pregnant patients with a clinical diagnosis of preeclampsia with severe features
  * gestational age between 23+0 and 32+0 weeks' gestation
  * singleton pregnancy
  * age 18-50 years old
  * No indication for immediate delivery (e.g. the patient and their physician team have planned expectant management of preeclampsia with severe features
  * Able to consent and follow a 2-step commend
  * English speaking
* Outpatient Cohort

  * Pregnant patients with a clinical diagnosis of preeclampsia without severe features
  * gestational age between 23+0 and 34+0 weeks' gestation
  * singleton pregnancy
  * age 18-50 years old
  * No indication for immediate delivery
  * Planned outpatient management of preeclampsia
  * Able to consent and follow a 2-step commend
  * English speaking

Exclusion Criteria:

* • Unable to stand from chair without physical assistance from another person (able to use assistive device).

  * History of blood clots in the extremities or any condition in which compression of the thigh or transient ischemia is contraindicated (i.e., wounds in the leg).
  * Chronic lasting symptoms (> 6 months) of severe COVID-19 (i.e., hospitalization)
  * History of head trauma or concussion within the past 6 months
  * Comorbid neurological disorder
  * Peripheral vascular disease
  * Diagnosed myocardial infarction or arrhythmia in the previous year
  * Resting SBP ≥180 mmHg or DBP ≥ 100 mmHg
  * Other significant medical condition likely to influence study or jeopardize safety as assessed by the Primary Investigator

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only patients who are pregnant are able to participate.
Enrollment: 80 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Brachial Artery Flow Mediated Dilation (FMD) | 1-2 times per week from enrollment until delivery, up to 10 months
  We will measure brachial artery vascular health in the arm. Baseline brachial artery diameter and blood flow velocity through the artery will be measured before and after a pneumatic forearm cuff is inflated to 225 mmHg for five minutes.

SECONDARY OUTCOMES:
Cutaneous Microvascular Function | 1-2 times per week From enrollment until delivery, up to to months.
  Laser Doppler Flowmetry (LDF) will measure blood flow flux during local skin heating to examine microvessel vasodilation
Placental Microvascular Function | At Delivery
  After delivery, placental vessels will be isolated from the placenta and a videomicroscopy technique will be used to evaluate flow-mediated dilation in vessels from placebo and MitoQ treated pregnancies.
Time from Enrollment to Delivery | Time in days from enrollment to delivery, up to 10 months
  Time from diagnosis and initiation of MitoQ or placebo to delivery
Blood Draw | Weekly from enrollment until Delivery, up to 10 months
  We will collect blood each week. The blood draw analysis may include but will not be limited to examining sFlt:PlGF ratio, plasma redox and bioenergetic analyses.
Maternal Preeclampsia Severity | From enrollment until delivery, up to 10 months
  A composite outcome of Maternal Severity of preeclampsia will be assessed and include laboratory, blood pressure, and ultrasound data relevant to preeclampsia
Composite Neonatal Delivery Outcome | Collected from delivery until hospital discharge; up to 1 week after birth.
  A composite outcome of neonatal delivery information including (but not limited to): cord blood, gestational age, weight, APGARs

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer J McIntosh, D.O.,, Principal Investigator — Medical College of Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
The cleaned, item-level spreadsheet data for all variables will be shared openly, along with example quantifications and transformations from initial raw data. Final files used to generate specific analyses as well as related results will also be shared. The rationale for sharing only cleaned data is to foster ease of data reuse. The final dataset will include clinical data procured from demographic and relevant medical record information from participants. We will share de-identified individual-participant level (IPD) data. Appropriate de-identification measures will be utilized from IRB approved protocols and informed consents.
Time Frame: Data will be made available 2 years after the completion of the study.
Access Criteria: Those interested in accessing the data will contact the PI and the study team will review requests and share relevant de-identified individual-participant level (IPD) data .

REFERENCES:
- [Background] Vangrieken P, Al-Nasiry S, Bast A, Leermakers PA, Tulen CBM, Schiffers PMH, van Schooten FJ, Remels AHV. Placental Mitochondrial Abnormalities in Preeclampsia. Reprod Sci. 2021 Aug;28(8):2186-2199. doi: 10.1007/s43032-021-00464-y. Epub 2021 Feb 1. PMID 33523425
- [Background] Chekir C, Nakatsuka M, Noguchi S, Konishi H, Kamada Y, Sasaki A, Hao L, Hiramatsu Y. Accumulation of advanced glycation end products in women with preeclampsia: possible involvement of placental oxidative and nitrative stress. Placenta. 2006 Feb-Mar;27(2-3):225-33. doi: 10.1016/j.placenta.2005.02.016. Epub 2005 Apr 22. PMID 16338468
- [Background] Zsengeller ZK, Rajakumar A, Hunter JT, Salahuddin S, Rana S, Stillman IE, Ananth Karumanchi S. Trophoblast mitochondrial function is impaired in preeclampsia and correlates negatively with the expression of soluble fms-like tyrosine kinase 1. Pregnancy Hypertens. 2016 Oct;6(4):313-319. doi: 10.1016/j.preghy.2016.06.004. Epub 2016 Jun 30. PMID 27939475
- [Background] Opichka MA, Livergood MC, Balapattabi K, Ritter ML, Brozoski DT, Wackman KK, Lu KT, Kozak KN, Wells C, Fogo AB, Gibson-Corley KN, Kwitek AE, Sigmund CD, McIntosh JJ, Grobe JL. Mitochondrial-targeted antioxidant attenuates preeclampsia-like phenotypes induced by syncytiotrophoblast-specific Galphaq signaling. Sci Adv. 2023 Dec;9(48):eadg8118. doi: 10.1126/sciadv.adg8118. Epub 2023 Dec 1. PMID 38039359
- [Background] Oyewole AO, Birch-Machin MA. Mitochondria-targeted antioxidants. FASEB J. 2015 Dec;29(12):4766-71. doi: 10.1096/fj.15-275404. Epub 2015 Aug 7. PMID 26253366
- [Background] Vaka R, Deer E, LaMarca B. Is Mitochondrial Oxidative Stress a Viable Therapeutic Target in Preeclampsia? Antioxidants (Basel). 2022 Jan 22;11(2):210. doi: 10.3390/antiox11020210. PMID 35204094
- [Background] Teran E, Hernandez I, Nieto B, Tavara R, Ocampo JE, Calle A. Coenzyme Q10 supplementation during pregnancy reduces the risk of pre-eclampsia. Int J Gynaecol Obstet. 2009 Apr;105(1):43-5. doi: 10.1016/j.ijgo.2008.11.033. Epub 2009 Jan 19. PMID 19154996
- [Background] Weissgerber TL, Milic NM, Milin-Lazovic JS, Garovic VD. Impaired Flow-Mediated Dilation Before, During, and After Preeclampsia: A Systematic Review and Meta-Analysis. Hypertension. 2016 Feb;67(2):415-23. doi: 10.1161/HYPERTENSIONAHA.115.06554. Epub 2015 Dec 28. PMID 26711737
- [Background] Stanhewicz AE, Nuckols VR, Pierce GL. Maternal microvascular dysfunction during preeclamptic pregnancy. Clin Sci (Lond). 2021 May 14;135(9):1083-1101. doi: 10.1042/CS20200894. PMID 33960392
- [Background] Sanchez-Aranguren LC, Prada CE, Riano-Medina CE, Lopez M. Endothelial dysfunction and preeclampsia: role of oxidative stress. Front Physiol. 2014 Oct 10;5:372. doi: 10.3389/fphys.2014.00372. eCollection 2014. PMID 25346691